CLINICAL TRIAL: NCT00132587
Title: Prospective Randomized Study of 130 Total Knee Arthroplasty With Cemented Femoral Implant Versus Cementless
Brief Title: Total Knee Arthroplasty (TKA) Cemented Versus Cementless
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Philippe Neyret, Hospices Civils de Lyon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2003.313
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2008-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee arthroplasty; Femoral loosening; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

INTERVENTIONS:
Device: cement Palacos R40 and LV40

SUMMARY:
The aim of the study is to analyse and to compare the quality of fixation of a femoral implant with or without cement.

One hundred thirty patients will be operated on and included with 2 groups, the first one with TKA all cemented and the second one with TKA with a cementless femoral implant. The study criteria include the IKS (International Knee Society) score and the analysis of a radiolucent line at the femur.

Patients will be reviewed at 2, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis (medial and/or lateral femoro-tibial arthritis and/or patellofemoral arthritis)
* Indication of surgical treatment by total knee arthroplasty
* Age between 50 and 90 years
* Acceptance and signature to participate

Exclusion Criteria:

* Rheumatoid or other inflammatory arthritis
* Association with other surgical procedure (osteotomy)
* Range of motion inferior to 90°
* Previous knee surgery (except arthroscopy)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2004-03; Primary Completion 2006-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
IKS (International Knee Society) score at 12 months

SECONDARY OUTCOMES:
Analysis of femoral radiolucent line at the X-rays (profile and anterior-posterior [AP] view) at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe NEYRET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix-Rousse, Lyon, France

REFERENCES:
- [Result] Demey G, Servien E, Pinaroli A, Lustig S, Ait Si Selmi T, Neyret P. The influence of femoral cementing on perioperative blood loss in total knee arthroplasty: a prospective randomized study. J Bone Joint Surg Am. 2010 Mar;92(3):536-41. doi: 10.2106/JBJS.H.01159. PMID 20194310